CLINICAL TRIAL: NCT03105505
Title: The Efficacy Of Lyclear (Permethrin 5%) Vs Fusidic Acid1% and Synthomycine 5% for Demodex -Blepharitis Treatment, Prospective-Randomized Trial.
Brief Title: The Efficacy of Permethrin 5%, Fusidic Acid 1% and Synthomycine 5% for Demodex - Blepharitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Barzilai Medical Center (Other)
Responsible Party: Principal Investigator, Igor Kaiserman, Prof Igor Kaiserman, Barzilai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 003-16-BRZ
Record Dates: First submitted 2017-03-28; First posted 2017-04-10 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Inflammation of the Eyelids
MeSH Terms: interventions — Fusidic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Permethrin 5% (Active Comparator): Contains permethrin 5% w/w (equivalent to 50 mg/g), formaldehyde solution 0.278% w/w and butylated hydroxytoluene (E321) 0.02% w/w.
  Interventions: Drug: Permethrin 5%
- Synthomycine 5%, (Active Comparator): Contains chloramphenicol 5%.
  Interventions: Drug: Synthomycine 5%
- Fusidic Acid 1% (Active Comparator): Contains 1% w/w fusidic acid anhydrous (as the hemihydrates) and 0.011% w/w.
  Interventions: Drug: Fusidic Acid 1% M/R Eye Drops

INTERVENTIONS:
Drug: Permethrin 5% — Facial skin application once a night for 3 months.
  Arms: Permethrin 5%
Drug: Synthomycine 5% — Eye ointment, eyelids and eyelashes application (chloramphenicol), once a night for 3 months.
  Arms: Synthomycine 5%,
Drug: Fusidic Acid 1% M/R Eye Drops — viscous eye drops application once a night for 3 months.
  Arms: Fusidic Acid 1%

SUMMARY:
The study aims to investigate the effect of Permethrin 5% treatment on Signs and symptoms of Demodex-blepharitis in comparison to Synthomycine 5% and Fucithalmic (fusidic acid 1%) .

DETAILED DESCRIPTION:
3 arms study. 75 patient total, 25 patients in each group.

Group A (study group) patients will apply facially Permethrin 5% every night for 3 months.

Group B patients will apply on the eyelids Fusidic acid 1% every night for 3 months.

Group C patients will apply on the eyelids Synthomycine 5% every night for 3 months

Follow up Evaluation will be made after one week, one month, two months, three months, 4 months and half a year.

ELIGIBILITY:
Inclusion Criteria:

- Adult (Age ≥18Y) individuals clinically diagnosed with Demodex- blepharitis.

Exclusion Criteria:

- Known sensitivity to all study medications or components. Pregnant women and individuals deemed unfit to provide informed consent. Systemic steroid use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Decrease in demodex infestation in group A (permethrin 5%). | 2 months
  significant decrease in demodex infestation in comparison to group B and C.
Improvement in symptoms and complaints in group A. | 2 months
  OSDI Questionnaires that describe the severity of the ocular surface disease condition are filled in each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Barzilai Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: Undecided